CLINICAL TRIAL: NCT01476475
Title: A Randomized, 24-week, Open-label, 2-arm Parallel-group, Multicenter Study Comparing the Efficacy and Safety of Insulin Glargine/Lixisenatide Fixed Ratio Combination Versus Insulin Glargine on Top of Metformin in Type 2 Diabetic Patients
Brief Title: Efficacy and Safety of Insulin Glargine/Lixisenatide Fixed Combination Versus Insulin Glargine Alone on Top of Metformin in Type 2 Diabetic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACT12374; 2011-002090-36 (EudraCT Number); U1111-1121-7111 (Other: UTN)
Record Dates: First submitted 2011-11-04; First posted 2011-11-22 (Estimated); Results first posted 2017-02-10 (Actual); Last update posted 2017-02-10 (Actual); Status verified 2016-12

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; lixisenatide; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Insulin glargine/Lixisenatide Fixed Ratio Combination (FRC) (Experimental): FRC injected once daily (QD) for 24 weeks. Dose individually adjusted.
  Interventions: Drug: Insulin glargine /lixisenatide Fixed Ratio Combination; Drug: Metformin (Background drug)
- Insulin glargine (Active Comparator): Insulin glargine QD for 24 weeks. Dose individually adjusted.
  Interventions: Drug: Insulin glargine; Drug: Metformin (Background drug)

INTERVENTIONS:
Drug: Insulin glargine /lixisenatide Fixed Ratio Combination — FRC was self-administered by subcutaneous (SC) injection within 1 hour before breakfast using pen-type injector (Tactipen®): 100 U/ml insulin glargine and 50 mcg Lixisenatide (ratio of 2 U/1 mcg). The initial dose was 10 U/5 mcg and then dose was adjusted weekly to reach and maintain fasting self-monitored plasma glucose (SMPG) of 80 mg/dL to 100 mg/dL (4.4 mmol/L to 5.6 mmol/L.
  Other Names: (HOE901/AVE0010)
  Arms: Insulin glargine/Lixisenatide Fixed Ratio Combination (FRC)
Drug: Insulin glargine — Insulin glargine (100 U/ml) was self-administered by SC injection before breakfast using pen-type injector (Lantus® Solostar®). The initial daily dose of insulin glargine was 10 U and then dose was adjusted weekly to reach and maintain fasting SMPG of 80 mg/dL to 100 mg/dL (4.4 mmol/L to 5.6 mmol/L).
  Other Names: Lantus
  Arms: Insulin glargine
Drug: Metformin (Background drug) — Pharmaceutical form: Tablet; Route of administration: oral administration. To be kept at stable dose (≥1.5 g/day) throughout the study.

SUMMARY:
Primary Objective:

* The purpose of this study was to compare insulin glargine/ lixisenatide fixed ratio combination (FRC) versus insulin glargine on glycemic control over 24 weeks, as evaluated by glycosylated hemoglobin (HbA1c) reduction in type 2 diabetic participants treated with metformin.

Secondary Objectives:

* To compare insulin glargine/lixisenatide FRC versus insulin glargine over 24 weeks on:

  * Glycemic control in relation to a meal as evaluated by post-prandial plasma glucose and glucose excursions during a standardized meal test;
  * Percentage of participants reaching HbA1c <7% or ≤6.5%;
  * 7-point Self-Monitored Plasma Glucose (SMPG) profile;
  * Body weight;
  * Insulin glargine dose
  * Fasting Plasma Glucose (FPG);
  * Percentage of participants requiring rescue therapy during the 24-week open label treatment period;
* To assess safety and tolerability of insulin glargine/lixisenatide FRC.

DETAILED DESCRIPTION:
Approximately 27 weeks including a 24-week treatment period.

ELIGIBILITY:
Inclusion criteria:

* Participants with type 2 diabetes mellitus diagnosed for at least 1 year.
* Metformin treatment at a stable dose of at least 1.5 g/day for at least 3 months prior to screening.

Exclusion criteria:

* Age < legal age of adulthood (18 years).
* Screening HbA1c <7% or >10%.
* Screening FPG >250 mg/dL (>13.9 mmol/L).
* Pregnancy or lactation, women of childbearing potential with no effective contraceptive method.
* Type 1 diabetes mellitus.
* Treatment with glucose-lowering agent(s) other than metformin in a period of 3 months prior to screening.
* Use of insulin within the last 6 months.
* Previous use of insulin, except for episode(s) of short-term treatment (≤15 consecutive days) due to intercurrent illness.
* Amylase and/or lipase >3 times the upper limit of the normal laboratory range (ULN) at screening.
* Calcitonin ≥20 pg/ml (5.9 pmol/l) at screening.
* Alanine Transferase (ALT) >3 ULN at screening.
* History of unexplained pancreatitis, chronic pancreatitis, pancreatectomy.
* Personal or immediate family history of medullary thyroid cancer (MTC) or genetic conditions that predisposes to MTC (e.g. multiple endocrine neoplasia syndromes).
* Uncontrolled or inadequately controlled hypertension at the time of screening with a resting supine systolic or diastolic blood pressure >180 mmHg or >110 mmHg, respectively.
* Within the last 6 months prior to screening: history of heart failure requiring hospitalization, myocardial infarction, or stroke. Planned coronary, carotid or peripheral artery revascularisation procedures.
* Body Mass Index (BMI) ≤20 or >40 kg/m^2.
* Any previous treatment with lixisenatide

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2011-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (70):
- United States (14):
  - Investigational Site Number 840408, Little Rock, Arkansas
  - Investigational Site Number 840412, Paramount, California
  - Investigational Site Number 840401, Larenceville, Georgia
  - Investigational Site Number 840417, Roswell, Georgia
  - Investigational Site Number 840403, Lexington, Kentucky
  - Investigational Site Number 840404, Hyattsville, Maryland
  - Investigational Site Number 840405, Rockville, Maryland
  - Investigational Site Number 840411, Las Vegas, Nevada
  - Investigational Site Number 840415, West Seneca, New York
  - Investigational Site Number 840402, Norman, Oklahoma
  - Investigational Site Number 840407, Medford, Oregon
  - Investigational Site Number 840413, Durham, Pennsylvania
  - Investigational Site Number 840410, Dallas, Texas
  - Investigational Site Number 840414, Renton, Washington
- Chile (5):
  - Investigational Site Number 152404, Santiago
  - Investigational Site Number 152405, Santiago
  - Investigational Site Number 152403, Santiago
  - Investigational Site Number 152401, Santiago
  - Investigational Site Number 152402, Santiago
- Czechia (4):
  - Investigational Site Number 203403, Nový Jičín
  - Investigational Site Number 203401, Pilsen
  - Investigational Site Number 203402, Prague
  - Investigational Site Number 203405, Prague
- Denmark (4):
  - Investigational Site Number 208401, København NV
  - Investigational Site Number 208404, Køge
  - Investigational Site Number 208402, Slagelse
  - Investigational Site Number 208403, Svendborg
- France (3):
  - Investigational Site Number 250402, Narbonne
  - Investigational Site Number 250404, Poitiers
  - Investigational Site Number 250401, Vandœuvre-lès-Nancy
- Germany (3):
  - Investigational Site Number 276401, Dresden
  - Investigational Site Number 276402, Ludwigshafen
  - Investigational Site Number 276403, Oberhausen
- Hungary (6):
  - Investigational Site Number 348401, Balatonfüred
  - Investigational Site Number 348405, Budapest
  - Investigational Site Number 348406, Budapest
  - Investigational Site Number 348404, Debrecen
  - Investigational Site Number 348402, Szeged
  - Investigational Site Number 348403, Szeged
- Lithuania (4):
  - Investigational Site Number 440401, Kaunas
  - Investigational Site Number 440402, Kaunas
  - Investigational Site Number 440403, Kėdainiai
  - Investigational Site Number 440404, Klaipėda
- Mexico (5):
  - Investigational Site Number 484404, Acapulco
  - Investigational Site Number 484401, Cuernavaca
  - Investigational Site Number 484405, Durango
  - Investigational Site Number 484402, Guadalajara
  - Investigational Site Number 484403, Guadalajara
- Poland (7):
  - Investigational Site Number 616405, Bialystok
  - Investigational Site Number 616406, Gdansk
  - Investigational Site Number 616403, Krakow
  - Investigational Site Number 616407, Lodz
  - Investigational Site Number 616404, Puławy
  - Investigational Site Number 616402, Szczecin
  - Investigational Site Number 616401, Warsaw
- Romania (6):
  - Investigational Site Number 642402, Brasov
  - Investigational Site Number 642403, Bucharest
  - Investigational Site Number 642405, Iași
  - Investigational Site Number 642401, Oradea
  - Investigational Site Number 642406, Târgu Mureş
  - Investigational Site Number 642404, Timișoara
- Slovakia (6):
  - Investigational Site Number 703402, Bratislava
  - Investigational Site Number 703403, Košice
  - Investigational Site Number 703406, Košice
  - Investigational Site Number 703404, Moldava nad Bodvou
  - Investigational Site Number 703405, Nitra
  - Investigational Site Number 703401, Žilina
- Sweden (3):
  - Investigational Site Number 752402, Skellefteå
  - Investigational Site Number 752401, Stockholm
  - Investigational Site Number 752403, Vaxjo

REFERENCES:
- [Result] Rosenstock J, Diamant M, Aroda VR, Silvestre L, Souhami E, Zhou T, Perfetti R, Fonseca V; LixiLan PoC Study Group. Efficacy and Safety of LixiLan, a Titratable Fixed-Ratio Combination of Lixisenatide and Insulin Glargine, Versus Insulin Glargine in Type 2 Diabetes Inadequately Controlled on Metformin Monotherapy: The LixiLan Proof-of-Concept Randomized Trial. Diabetes Care. 2016 Sep;39(9):1579-86. doi: 10.2337/dc16-0046. Epub 2016 Jun 9. PMID 27284114
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pubmed/?term=27284114

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 70 centers in 13 countries. A total of 520 participants were screened between November 21, 2011 and June 08, 2012. Out of 520 participants, 197 were screen failure; main reason for screen failure was that glycosylated hemoglobin (HbA1c) values were out of the protocol defined range.
Pre-assignment Details: A total of 323 participants were randomized in 1:1 ratio to insulin glargine/lixisenatide fixed ratio combination (FRC) and insulin glargine arms, stratified by screening HbA1c values (<8% or ≥8%) and screening body mass index (BMI) values (<30 kg/m^2, ≥30 kg/m^2).
Groups:
- Insulin Glargine/Lixisenatide Fixed Ratio Combination: FRC injected subcutaneously once daily (QD) for 24 weeks. Dose individually adjusted.
- Insulin Glargine: Insulin glargine injected subcutaneously QD for 24 weeks. Dose individually adjusted.
Period: Overall Study
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination | Insulin Glargine
Started | 161 | 162
Completed | 150 | 159
Not Completed | 11 | 3
Not completed — Adverse Event | 6 | 0
Not completed — Poor compliance to protocol | 1 | 1
Not completed — Other reasons | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Insulin Glargine/Lixisenatide Fixed Ratio Combination: FRC injected subcutaneously QD for 24 weeks. Dose individually adjusted.
- Total: Total of all reporting groups
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination | Insulin Glargine | Total
Number analyzed (Participants) | 161 | 162 | 323
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.9 (9.5) | 56.6 (9.4) | 56.7 (9.4)
Gender [Count of Participants; unit: Participants]
  Female | 81 | 77 | 158
  Male | 80 | 85 | 165
Race [Number; unit: participants]
  Caucasian/White | 158 | 160 | 318
  Black | 2 | 1 | 3
  Asian/Oriental | 1 | 1 | 2
Ethnicity [Number; unit: participants]
  Hispanic | 35 | 30 | 65
  Non Hispanic | 126 | 132 | 258
Screening HbA1c [Mean (Standard Deviation); unit: percentage of haemoglobin] | 8.12 (0.80) | 8.08 (0.77) | 8.10 (0.78)
Baseline BMI [Mean (Standard Deviation); unit: kg/m^2] | 32.24 (4.75) | 32.02 (4.35) | 32.13 (4.55)
Duration of Diabetes [Mean (Standard Deviation); unit: years] | 6.29 (4.29) | 7.10 (5.27) | 6.69 (4.82)
Daily Dose of Metformin [Mean (Standard Deviation); unit: mg] | 2075.8 (440.7) | 2093.7 (415.5) | 2084.8 (427.7)
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] | 9.76 (2.19) | 9.46 (2.16) | 9.61 (2.18)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline to Week 24
Description: Change in HbA1c was calculated by subtracting baseline value from Week 24 value. Missing data was imputed using last observation carried forward (LOCF). On-treatment period for this efficacy variable was defined as the time from the first dose of study drug till before the introduction of rescue medication and up to 14 days after the last injection of investigational medicinal product (IMP).
Time Frame: Baseline, Week 24
Population: Modified intent-to-treat (mITT) population consisted of all randomized participants received at least 1 dose of IMP and had both baseline and at least 1 post-baseline efficacy assessment. Number of participants analyzed = participants with both baseline and at least one post-baseline HbA1c assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: percentage of hemoglobin
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination | Insulin Glargine
Number analyzed (Participants) | 160 | 161
percentage of hemoglobin | -1.82 (0.058) | -1.64 (0.057)
Statistical Analysis 1: Comparison: Insulin Glargine/Lixisenatide Fixed Ratio Combination vs Insulin Glargine; Analysis was performed using analysis of covariance (ANCOVA) model with treatment groups, randomization strata of screening HbA1c (<8.0, ≥8.0%), randomization strata of screening BMI (<30 kg/m^2, ≥30 kg/m^2), and country as fixed effects and baseline HbA1c value as covariates. A step-down testing procedure described by Hochberg and Tamhane was used to control type-1 error; Test type: Non-Inferiority or Equivalence — The non-inferiority of insulin glargine/lixisenatide FRC versus insulin glargine was tested first, at alpha level of 0.025 (1-sided) and a non-inferiority margin of 0.4% HbA1c. If non-inferiority was established, then a test of superiority of insulin glargine/lixisenatide FRC over insulin glargine would be performed, at alpha level of 0.05 (2-sided). The non-inferiority was assessed using upper bound of 2-sided 95% confidence interval (CI) at ≤0.4%; ANCOVA; Least square (LS) mean difference = -0.17, 95% CI 2-sided [-0.312 to -0.037], Standard Error of Mean 0.070 — Insulin glargine/Lixisenatide FRC vs Insulin glargine
Statistical Analysis 2: Comparison: Insulin Glargine/Lixisenatide Fixed Ratio Combination vs Insulin Glargine; Analysis was performed using ANCOVA model with treatment groups, randomization strata of screening HbA1c (<8.0, ≥8.0%), randomization strata of screening BMI (<30 kg/m^2, ≥30 kg/m^2), and country as fixed effects and baseline HbA1c value as covariates. If non-inferiority was established, then a test of superiority of insulin glargine/lixisenatide FRC over insulin glargine would be performed, at alpha level of 0.05 (2-sided); Test type: Superiority or Other; p = 0.0130, ANCOVA — Threshold for significance at 0.05 level; LS Mean Difference = -0.17, 95% CI 2-sided [-0.312 to -0.037], Standard Error of Mean 0.070 — Insulin glargine/Lixisenatide FRC vs Insulin glargine

2. Secondary Outcome: Change in 2-hour Postprandial Plasma Glucose (PPG) From Baseline to Week 24
Description: The 2-hour PPG test measured blood glucose 2 hours after eating a standardized meal. Change in PPG was calculated by subtracting baseline value from Week 24 value. Missing data was imputed using LOCF. On-treatment period for this efficacy variable was defined as the time from the first dose of study drug till before the introduction of rescue medication and up to the date of last injection of IMP.
Time Frame: Baseline, Week 24
Population: mITT population.Here, number of participants analyzed = participants with both baseline and at least one post-baseline 2-hour PPG assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination | Insulin Glargine
Number analyzed (Participants) | 151 | 153
mmol/L | -7.49 (0.283) | -4.33 (0.274)
Statistical Analysis 1: Comparison: Insulin Glargine/Lixisenatide Fixed Ratio Combination vs Insulin Glargine; Analysis was performed using ANCOVA with treatment groups,randomization strata of screening HbA1c(<8.0, ≥8.0%)& screening BMI(<30 kg/m^2, ≥30 kg/m^2),country as fixed effects and baseline 2-hour PPG value as covariates.A step-down testing procedure used to control type-1 error.If non-inferiority demonstrated for primary endpoint,superiority testing on secondary endpoints was performed sequentially in order endpoints are reported(continued only if previous endpoint was statistically significant); Test type: Superiority or Other; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; LS Mean Difference = -3.17, 95% CI 2-sided [-3.832 to -2.504], Standard Error of Mean 0.337 — Insulin glargine/Lixisenatide FRC vs Insulin glargine

3. Secondary Outcome: Change in 2-hour Plasma Glucose Excursion From Baseline to Week 24
Description: 2-hour plasma glucose excursion = 2-hour PPG minus plasma glucose value obtained 30 minutes prior to the start of the meal and before IMP administration. Change in plasma glucose excursion was calculated by subtracting baseline value from Week 24 value. Missing data was imputed using LOCF. On-treatment period for this efficacy variable was defined as the time from the first dose of study drug till before the introduction of rescue medication and up to the date of last injection of IMP.
Time Frame: Baseline, Week 24
Population: mITT population. Here, number of participants analyzed = participants with both baseline and at least one post-baseline plasma glucose excursion assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination | Insulin Glargine
Number analyzed (Participants) | 151 | 152
mmol/L | -3.91 (0.277) | -0.67 (0.269)
Statistical Analysis 1: Comparison: Insulin Glargine/Lixisenatide Fixed Ratio Combination vs Insulin Glargine; Testing according to the step-down testing procedure (continued only if previous endpoint was statistically significant). Analysis was performed using ANCOVA model with treatment groups, randomization strata of screening HbA1c (<8.0, ≥8.0%), randomization strata of screening BMI (<30 kg/m^2, ≥30 kg/m^2), and country as fixed effects and baseline 2-hour plasma glucose excursion value as covariates; Test type: Superiority or Other; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; LS Mean Difference = -3.24, 95% CI 2-sided [-3.895 to -2.592], Standard Error of Mean 0.331 — Insulin glargine/Lixisenatide FRC vs Insulin glargine

4. Secondary Outcome: Change in Average 7-Point Self-Monitored Plasma Glucose (SMPG) Profiles From Baseline to Week 24
Description: Participants recorded a 7-point plasma glucose profile measured before and 2-hours after each meal and at bedtime, over a single day, once in a week before baseline, before visit Week 12 and before visit Week 24 and the average value across the profiles performed in the week before a visit for the 7-time points was calculated. Change in average 7-point SMPG was calculated by subtracting baseline value from Week 24 value. Missing data was imputed using LOCF. On-treatment period for this efficacy variable was defined as the time from the first dose of study drug till before the introduction of rescue medication and up to the date of last injection of IMP.
Time Frame: Baseline, Week 24
Population: mITT population. Here, number of participants analyzed = participants with baseline and at least one post-baseline 7-point SMPG assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination | Insulin Glargine
Number analyzed (Participants) | 149 | 155
mmol/L | -3.23 (0.104) | -2.93 (0.101)
Statistical Analysis 1: Comparison: Insulin Glargine/Lixisenatide Fixed Ratio Combination vs Insulin Glargine; Testing according to the step-down testing procedure (continued only if previous endpoint was statistically significant). Analysis was performed using ANCOVA model with treatment groups, randomization strata of screening HbA1c (<8.0, ≥8.0%), randomization strata of screening BMI (<30 kg/m^2, ≥30 kg/m^2), and country as fixed effects and baseline average 7-point SMPG value as covariates; Test type: Superiority or Other; p = 0.0154, ANCOVA — Threshold for significance at 0.05 level; LS Mean Difference = -0.30, 95% CI 2-sided [-0.550 to -0.058], Standard Error of Mean 0.125 — Insulin glargine/Lixisenatide FRC vs Insulin glargine

5. Secondary Outcome: Change in Body Weight From Baseline to Week 24
Description: Change in body weight was calculated by subtracting baseline value from Week 24 value. Missing data was imputed using LOCF. On-treatment period for this efficacy variable was defined as the time from the first dose of study drug till before the introduction of rescue medication and up to 3 days after the last injection of IMP.
Time Frame: Baseline, Week 24
Population: mITT population. Here, number of participants analyzed = participants with baseline and at least one post-baseline body weight assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination | Insulin Glargine
Number analyzed (Participants) | 159 | 160
kg | -0.97 (0.289) | 0.48 (0.282)
Statistical Analysis 1: Comparison: Insulin Glargine/Lixisenatide Fixed Ratio Combination vs Insulin Glargine; Testing according to the step-down testing procedure (continued only if previous endpoint was statistically significant). Analysis was performed using ANCOVA model with treatment groups, randomization strata of screening HbA1c (<8.0, ≥8.0%), randomization strata of screening BMI (<30 kg/m^2, ≥30 kg/m^2), and country as fixed effects and baseline body weight value as covariates; Test type: Superiority or Other; p < 0.0001, ANCOVA — Threshold for significance at 0.05 level; LS Mean Difference = -1.44, 95% CI 2-sided [-2.110 to -0.773], Standard Error of Mean 0.340 — Insulin glargine/Lixisenatide FRC vs Insulin glargine

6. Secondary Outcome: Average Daily Insulin Glargine Dose at Week 24
Description: Missing data was imputed using LOCF. On-treatment period for this efficacy variable was defined as the time from the first dose of study drug till before the introduction of rescue medication and up to the date of last injection of IMP.
Time Frame: Week 24
Population: mITT population. Here, number of participants analyzed = participants with insulin glargine dose measured during on-treatment period
Measure: Least Squares Mean (Standard Error); unit: Units (U)
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination | Insulin Glargine
Number analyzed (Participants) | 161 | 162
Units (U) | 36.08 (1.415) | 39.32 (1.384)
Statistical Analysis 1: Comparison: Insulin Glargine/Lixisenatide Fixed Ratio Combination vs Insulin Glargine; Testing according to the step-down testing procedure (continued only if previous endpoint was statistically significant). Analysis was performed using ANCOVA model with treatment groups, randomization strata of screening HbA1c (<8.0, ≥8.0%), randomization strata of screening BMI (<30 kg/m^2, ≥30 kg/m^2), and country as fixed effects; Test type: Superiority or Other; p = 0.0583, ANCOVA — Threshold for significance at 0.05 level; LS Mean Difference = -3.24, 95% CI 2-sided [-6.592 to 0.114], Standard Error of Mean 1.704 — Insulin glargine/Lixisenatide FRC vs Insulin glargine

7. Secondary Outcome: Change in FPG From Baseline to Week 24
Description: Change in FPG was calculated by subtracting baseline value from Week 24 value. Missing data was imputed using LOCF. On-treatment period for this efficacy variable was defined as the time from the first dose of study drug till before the introduction of rescue medication and up to 1 day after the last injection of IMP.
Time Frame: Baseline, Week 24
Population: mITT population. Here, number of participants analyzed = participants with baseline and at least one post-baseline FPG assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination | Insulin Glargine
Number analyzed (Participants) | 159 | 160
mmol/L | -3.35 (0.130) | -3.51 (0.128)

8. Secondary Outcome: Percentage of Participants Requiring Rescue Therapy During 24-week Treatment Period
Description: Routine fasting SMPG and central laboratory FPG (and HbA1c after Week 12) values were used to determine the requirement of rescue medication. If fasting SMPG value exceed the specified limit for 3 consecutive days, the central laboratory FPG (and HbA1c after Week 12) were performed. Threshold values from Week 8 to Week 12: fasting SMPG/FPG >240 mg/dL (13.3 mmol/L), and from Week 12 to Week 30: fasting SMPG/FPG >200 mg/dL (11.1 mmol/L) or HbA1c >8%.
Time Frame: Baseline up to Week 24
Population: mITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination | Insulin Glargine
Number analyzed (Participants) | 161 | 162
percentage of participants | 0 | 0.6

9. Secondary Outcome: Percentage of Participants With HbA1c ≤6.5 % or <7.0 % at Week 24
Description: On-treatment period for this efficacy variable was defined as the time from the first dose of study drug till before the introduction of rescue medication and up to 14 days after the last injection of IMP.
Time Frame: Week 24
Population: mITT population. Here, number of participants analyzed = participants with at least one post-baseline HbA1c assessment during on-treatment period.
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination | Insulin Glargine
Number analyzed (Participants) | 160 | 161
percentage of participants
  HbA1c ≤6.5% | 71.9 | 64.6
  HbA1c <7.0% | 84.4 | 78.3

10. Secondary Outcome: Change in 30-minute and 1-hour PPG From Baseline to Week 24
Description: The 30 minute and 1-hour PPG test measured blood glucose 30 minutes and 1-hour after eating a standardized meal. Change in PPG was calculated by subtracting baseline value from Week 24 value. Missing data was imputed using LOCF. On-treatment period for this efficacy variable was defined as the time from the first dose of study drug till before the introduction of rescue medication and up to the date of last injection of IMP.
Time Frame: Baseline, Week 24
Population: mITT population. Here, number of participants analyzed = participants with baseline and at least one post-baseline PPG assessment during on-treatment period. Here, 'n' signifies number of participants with available data for specified category.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination | Insulin Glargine
Number analyzed (Participants) | 151 | 153
mmol/L
  30-minute PPG (n=151, 153) | -5.01 (0.194) | -3.76 (0.187)
  1-hour PPG (n=150, 153) | -5.94 (0.246) | -4.10 (0.239)

11. Secondary Outcome: Change in 30 Minute and 1-hour Plasma Glucose Excursion From Baseline to Week 24
Description: 30-minute and 1-hour plasma glucose excursion = 30-minute and 1-hour PPG minus plasma glucose value obtained 30 minutes prior to the start of the meal and before IMP administration. Change in plasma glucose excursion was calculated by subtracting baseline value from Week 24 value. Missing data was imputed using LOCF. On-treatment period for this efficacy variable was defined as the time from the first dose of study drug till before the introduction of rescue medication and up to the date of last injection of IMP.
Time Frame: Baseline, Week 24
Population: mITT population. Here, number of participants analyzed = participants with baseline and at least one post-baseline plasma glucose excursion assessment during on-treatment period.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination | Insulin Glargine
Number analyzed (Participants) | 151 | 152
mmol/L
  30-minute plasma glucose excursion (n=151, 152) | -1.47 (0.156) | -0.05 (0.151)
  1-hour plasma glucose excursion (n=150, 152) | -2.34 (0.233) | -0.44 (0.226)

12. Secondary Outcome: Percentage of Participants Reaching HbA1c <7% at Week 24 With no Documented Symptomatic Hypoglycemia During 24-week Treatment Period
Description: Documented symptomatic hypoglycemia was an event during which typical symptoms of hypoglycemia were accompanied by a measured plasma glucose concentration of ≤70 mg/dL (3.9 mmol/L). Participants without any post-baseline on-treatment value for HbA1c were counted as non-responders if they experienced at least one documented symptomatic hypoglycemia before the introduction of rescue medication and up to 1 day after the last injection of IMP. Otherwise, they were counted as missing data. On-treatment period for this efficacy variable was defined as the time from the first dose of study drug till before the introduction of rescue medication and up to 14 days after the last injection of IMP.
Time Frame: Baseline up to Week 24
Population: as for outcome 9
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination | Insulin Glargine
Number analyzed (Participants) | 160 | 161
percentage of participants | 67.5 | 59.0

13. Secondary Outcome: Percentage of Participants Reaching HbA1c <7% With no Body Weight Gain at Week 24
Description: Participants without any post-baseline on-treatment values (for HbA1c and body weight) that were no more than 30 days apart were counted as non-responders if at least one of the components (for HbA1c and body weight) was available and showed non-response. Otherwise, they were counted as missing data.
Time Frame: Week 24
Population: mITT population. Here, number of participants analyzed = participants with any post-baseline on-treatment values (for HbA1c and body weight) that were no more than 30 days apart or with one of the components (for HbA1c and body weight) showing non-response based on the last post-baseline on-treatment value.
Measure: Number; unit: percentage of participants
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination | Insulin Glargine
Number analyzed (Participants) | 160 | 161
percentage of participants | 56.3 | 37.3

14. Secondary Outcome: Percentage of Participants With Documented Symptomatic and Severe Symptomatic Hypoglycemia
Description: Documented symptomatic hypoglycemia was an event during which typical symptoms of hypoglycemia were accompanied by a measured plasma glucose concentration of ≤70 mg/dL (3.9 mmol/L).Severe symptomatic hypoglycemia was an event requiring assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions. These episodes were associated with sufficient neuroglycopenia to induce seizure, unconsciousness or coma. All episodes in which neurological impairment was severe enough to prevent self-treatment and which were thought to place participants at risk for injury to themselves or others.
Time Frame: First dose of study drug up to 3 days after the last dose administration (maximum of 219 days)
Population: Safety population that included all randomized participants who received at least 1 dose of study medication regardless of the amount of treatment administered.
Measure: Number; unit: percentage of participants
Groups:
- Insulin Glargine (Lantus® SoloSTAR®): Insulin glargine injected subcutaneously QD for 24 weeks. Dose individually adjusted.
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination | Insulin Glargine (Lantus® SoloSTAR®)
Number analyzed (Participants) | 161 | 162
percentage of participants
  Documented symptomatic hypoglycemia | 21.7 | 22.8
  Severe Symptomatic Hypoglycemia | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: All Adverse events (AEs) were collected from signature of the informed consent from up to the final visit (Week 24) regardless of seriousness or relationship to investigational product.
Description: Reported adverse events are treatment-emergent AEs that is AEs that developed/worsened during the 'on treatment period' (time from the first injection of open-label IMP up to 3 days after the last injection of IMP, regardless of the introduction of rescue therapy).
Groups:
- Insulin Glargine/Lixisenatide Fixed Ratio Combination: FRC injected subcutaneously QD for 24 weeks. Dose individually adjusted (median exposure: 169 days).
- Insulin Glargine: Insulin glargine injected subcutaneously QD for 24 weeks. Dose individually adjusted (median exposure: 169 days).
Arm/Group | Insulin Glargine/Lixisenatide Fixed Ratio Combination | Insulin Glargine
Serious Adverse Events (participants affected / at risk) | 9/161 | 6/162
Other Adverse Events (participants affected / at risk) | 26/161 | 21/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Insulin Glargine/Lixisenatide Fixed Ratio Combination (N=161) | Insulin Glargine (N=162)
Cellulitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Diabetic neuropathy (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 1 | 0
ECG signs of myocardial ischaemia (Investigations) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Insulin Glargine/Lixisenatide Fixed Ratio Combination (N=161) | Insulin Glargine (N=162)
Nasopharyngitis (Infections and infestations) | 9 | 9
Headache (Nervous system disorders) | 8 | 12
Nausea (Gastrointestinal disorders) | 12 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.